Official Title of the study: A Newly Modified Technique for Levator Muscle Tucking in

Blepharoptosis Surgery: An Egyptian tertiary center study

Date: 5/5/2021

**Study Protocol with SAP:** 

Background: To highlight a newly modified technique for levator muscle tucking for the management of

mild to moderate blepharoptosis.

**Methods**: A prospective single-centre study enrolling 180 patients with blepharoptosis at Ain Shams

University Hospitals from March 2017 to February 2019. Patients of unilateral or bilateral mild to moderate

ptosis with good levator function (more than 8 mm) were included. Those with severe, traumatic, recurrent,

mechanical ptosis, Marcus-Gunn jaw winking syndrome, third nerve palsy, absent Bell's phenomenon, or

abnormal ocular motility were excluded. The follow-up was at one week, one month, three months, six

months, and one year visits. Functional outcome was assessed by analysis of the upper eyelid margin

position in relation to the superior limbus and classified as very good (2 mm), good (2-4 mm), poor (5 mm)

and preoperative to postoperative difference in marginal reflex distance (MRD). The aesthetic outcome was

assessed in the form of symmetry of eyelid height, lid contour, lid crease presence, and degree of patient's

postoperative satisfaction.

Statistical analysis Plan:

Statistical analysis was performed using SPSS for Windows (version 22, SPSS, IBM Inc.). Pearson's chi-

square test was used to compare the values of preoperative and postoperative functional outcomes.

Descriptive statistics were used in the outcome. Statistical tests were performed at the 95% confidence

interval.